CLINICAL TRIAL: NCT06405685
Title: A Prospective, Single Arm Study of Nimotuzumab Combined With Gemcitabine and Nab-paclitaxel as Conversion Therapy in Pancreatic Cancer With Liver Metastasis
Brief Title: Nimotuzumab Plus AG in Pancreatic Cancer With Liver Metastasis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IST-Nim-PC-5
Record Dates: First submitted 2024-05-05; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2023-05

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — nimotuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nimotuzumab+AG (Experimental): Patients will receive Nimotuzumab plus AG as conversion therapy, and imaging assessments (according to RECIST V.1.1 criteria) will be performed every two cycles (every two months) of conversion therapy.
  Interventions: Drug: Nimotuzumab; Drug: AG

INTERVENTIONS:
Drug: Nimotuzumab — Nimotuzumab 400 mg will be administered on Day 1, 8, 15 of a 28-day cycle by intravenous (IV) administration up to 6 cycles. Imaging (CT or MRI) and tumor markers (such as CA19-9) will be assessed every two cycles of the conversion therapy, until met the criteria of resection and underwent surgery.
  Other Names: h-R3
Drug: AG — Patients will receive AG as conversion therapy up to 6 months. Gemcitabine 1000 mg/m^2 will be administered on Day 1, 8, 15 of a 28-day cycle. nab-Paclitaxel 125 mg/m^2 will be administered on Day 1, 8, 15 of a 28-day cycle by intravenous (IV) administration up to 6 cycles. Imaging (CT or MRI) and tumor markers (such as CA19-9) will be assessed every two cycles of the conversion therapy, until met the criteria of resection and underwent surgery.

SUMMARY:
This is a prospective, open-label, single arm clinical study. The main purpose of the study is to evaluate the clinical efficacy and safety of Nimotuzumab combined with AG in the treatment of pancreatic cancer with liver metastasis. Patients will receive Nimotuzumab plus AG as conversion therapy, and imaging assessments (according to RECIST V.1.1 criteria) will be performed every two cycles (every two months) of conversion therapy. The main endpoint is R0 resection rate. Additional end points included resection rates, overall survival (OS), objective response rate (ORR), safety, etc.

DETAILED DESCRIPTION:
This clinical study is designed as a prospective, open-label, single arm study to evaluate the clinical efficacy and safety of Nimotuzumab combined with AG (gemcitabine and nab-paclitaxel) in the treatment of pancreatic cancer with liver metastasis. Patients will receive Nimotuzumab plus AG as conversion therapy, and imaging assessments (according to RECIST V.1.1 criteria) will be performed every two cycles (every two months) of conversion therapy. The resectability of the primary pancreatic lesion and liver metastases will be judged based on NCCN guidelines and will be determined by a multidisciplinary team of experts. The main endpoint is R0 resection rate. Additional end points included resection rates, overall survival (OS), objective response rate (ORR), safety, etc.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 18-75 years old, gender unlimited;
* 2. Histologically or cytologically confirmed pancreatic cancer with liver metastasis;
* 3. Pancreatic cancer with liver metastasis, which is considered to be potentially resectable judged by a multidisciplinary team;
* 4. Receive nimotuzumab-based conversion therapy for voluntary;
* 5. No prior tumor systemic therapy;
* 6. Measurable disease according to RECIST criteria v1.1;
* 7. Adequate organ and bone marrow function, defined as follows: hemoglobin≥9.0 g/dL; absolute neutrophil count (ANC)≥1.5×10^9/L; platelets≥100×10^9/L; serum total bilirubin (TBIL)≤3×ULN; aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 5 times the upper limit of normal (ULN); serum creatinine≤1.5×ULN or estimated creatinine clearance > 60 mL/min;
* 8. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
* 9. Life expectancy is expected to be ≥3 months;
* 10. Fertile subjects are willing to take contraceptive measures during the study period.
* 11. Good compliance and signed informed consent voluntarily.

Exclusion Criteria:

* 1. Refuse chemotherapy or surgery;
* 2. Other part (e.g. peritoneum, lung, bone, brain) metastasis;
* 3. History of other malignancies (except cured basal cell carcinoma of the skin and carcinoma in situ of the cervix);
* 4. Accompanied by other serious diseases, including but not limited to: compensatory heart failure (NYHA grade III and IV), unstable angina, poorly controlled arrhythmias, uncontrolled hypertension (SBP>160mmHg or DBP>100mmHg); active infections; unmanageable diabetes mellitus; presence of uncontrolled pleural effusion, pericardial effusion, or ascites requiring drainage; severe portal hypertension; gastric outlet obstruction; Respiratory insufficiency;
* 5. Undergone major surgery within 30 days;
* 6. Use of EGFR-mab or EGFR-TKI within 30 days;
* 7. Known allergy to prescription or any component of the prescription used in this study;
* 8. With HIV, HPV, or syphilis infection, or active hepatitis (hepatitis B, hepatitis C);
* 9. Grade 2 or above toxicity from prior treatment that has not resolved (excluding anemia, alopecia, skin pigmentation, and chemotherapy-induced neurotoxicity)
* 10.Other reasons that are not suitable to participate in this study according to the researcher's judgment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-04-27 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
R0 resection rate | Up to 6 months
  The Proportion of patients who achieved R0 resection (incisal edge>1cm)

SECONDARY OUTCOMES:
resection rate | Up to 18 months
  The proportion of patients who underwent surgery.
overall survival (OS) | Up to 18 months
  The time from the beginning of treatment to death due to any cause.
Objective response rate (ORR) | Up to 18 months
  Objective response rate (ORR), including complete response (CR) and partial response (PR). Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT/MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), at least a 30% decrease in the sum of the longest diameter of target lesions.
tumor-related markers | Up to 18 months
  To explore the influence of tumor-related markers (such as CA199,EGFR) on prognosis.
adverse events | Up to 30 days after last administration
  Frequency and severity of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Jihui Hao, Dr, Study Chair — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No